CLINICAL TRIAL: NCT05359094
Title: To Explore the Effect of Probiotic Supplements in Chronic Kidney Disease
Brief Title: Probiotic Supplements in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SF22054A
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease
Keywords: Probiotics; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo
- Probiotics (Active Comparator): Probiotics
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo (Microcrystalline α-cellulose) supplement with a Plant-Dominant Low-Protein Diet
  Arms: Placebo
Dietary Supplement: Probiotics — Probiotics(Pediococcus acidilactici GKA4) supplement with a Plant-Dominant Low-Protein Diet
  Arms: Probiotics

SUMMARY:
This research will investigate the effect of oral probiotic supplements on renal function, uremic toxins inflammatory response, nutrition status, gastrointestinal symptoms, and QoL with Chronic kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) with gut microbiota was different from a normal person. Some gut microbiota produces short-chain fatty acids or induces functional enzymes beneficial to patients. On the other hand, some gut microbiota may also metabolize amino acids into p-cresol and indole which were leading to the accumulation of urinary toxins and damage to the kidney. This research will investigate the effect of oral probiotic supplements on renal function, uremic toxins, inflammatory response, nutrition status, gastrointestinal symptoms, and QoL with CKD.

ELIGIBILITY:
Inclusion criteria:

1. Aged over 20 years old.
2. Patients with 2~3a stage chronic kidney disease.
3. Those who can cooperate with the research plan for 3 visits and retain samples (blood, urine).

Exclusion criteria::

1. Use of other probiotics during the study.
2. Those with active infectious diseases in the past month.
3. Those who have used antibiotics within the past 1 month or during the study.
4. Women who are pregnant or breastfeeding.
5. Obstructive nephropathy within the past month.
6. Polycystic kidney disease (polycystic kidney disease).
7. Acute kidney disease within the past 3 months.
8. Gastrointestinal bleeding within the past 3 months.
9. Malignancy.
10. Severe cardiovascular disease (cardiovascular disease) in the past 3 months, such as coronary artery disease (coronary artery disease), myocardial ischemia (myocardial ischemia), NYHA class IV myocardial failure, cerebrovascular disease, or peripheral artery disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) measurement | Baseline to 24 week
  The eGFR level is a maker for kidney function
Blood Urea Nitrogen (BUN) levels | Baseline to 24 week
  Blood Urea Nitrogen
Electrolytes Analysis | Baseline to 24 week
  The concentration of electrolytes analysis in the subject's blood samples

SECONDARY OUTCOMES:
Uremic toxins assay | Baseline to 24 week
  The concentration of p-cresol sulfate level, indoxyl sulfates level, and trimethylamine N-oxide level (TMAO) in the subjects' blood samples
Sugar test | Baseline to 24 week
  The concentration of fasting sugar and HbA1C in the subjects' blood samples
Nutrition status | Baseline to 24 week
  The concentration of albumin,TIBC,TFS and uric acid in the subjects' blood samples
Inflammation makers | Baseline to 24 week
  The concentration of inflammation makers in the subjects' blood samples
Liver function | Baseline to 24 week
  The concentration of ALT and AST in the subjects' blood samples
Lipid analysis | Baseline to 24 week
  The concentration of total cholesterol , triglyceride , HDL-cholesterol and LDL-cholesterol in the subjects' blood samples
The quality of life | Baseline to 24 week
  Health-related quality of life was measured by 5-level EQ-5D questionnaire
Complete Blood Count (CBC) Test | Baseline to 24 week
  The concentration of CBC test in the subject's blood samples
Urine Analysis | Baseline to 24 week
  Urine specimen collection will be evaluate such as urine routine ,bacteria, protein and MCP-1.
24-hour Dietary recall | Baseline to 24 week
  There will be collected by food models or a photography atlas to estimate portion size.
Safety and compliance | Baseline to 24 week
  Gastrointestinal symptoms measured by questionnaire
Grip strength levels | Baseline to 24 week
  Hand grip strength was measured by grip strength device

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Chen, MDPHD, Principal Investigator — Division of Nephrology in Taichung Veterans General Hospital
Locations (1):
- Taiwan, Taichung, ROC, Taiwan